CLINICAL TRIAL: NCT04395222
Title: A Prospective Study of Tocilizumab for the Prevention of Graft Failure and Graft-versus-Host Disease in Haplo-Cord Transplantation
Brief Title: Tocilizumab for the Prevention of Graft Failure and GVHD in Haplo-Cord Transplantation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19-08020738
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Results first posted 2023-10-23 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Hematologic Malignancy; Bone Marrow Transplant
Keywords: Tocilizumab; Haplo-Cord Transplant; Allogeneic Transplant; Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — tocilizumab; fludarabine; fludarabine phosphate; Melphalan; Antilymphocyte Serum; thymoglobulin; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ATG Group I (Experimental): Anti-thymocyte Globulin (ATG) 1.5 mg/kg administered on Day -5, Day -3 and Day -1 of the transplant conditioning regimen.
  * Fludarabine 30mg/m2 administered on Day -7 through Day -3 of transplant conditioning regimen (if under 60 years old), or on Day -5 through Day -3 of transplant conditioning regimen (if over 60 years old)
  * Melphalan 140 mg/m2 administered on Day -2 of transplant conditioning regimen.
  * Total Body Irradiation 2 Gray administered on Day -4, Day -3 of transplant conditioning regimen.
  * Tocilizumab 8 mg/kg administered on Day -1 of transplant conditioning regimen.
  Interventions: Drug: Tocilizumab; Drug: Fludarabine; Drug: Melphalan; Drug: Anti-thymocyte globulin (rabbit); Radiation: Total Body Irradiation
- ATG Group II (Experimental): Anti-thymocyte Globulin (ATG) 1.5 mg/kg administered on Day -5, and Day -3 of the transplant conditioning regimen.
  * Fludarabine 30mg/m2 administered on Day -7 through Day -3 of transplant conditioning regimen (if under 60 years old), or on Day -5 through Day -3 of transplant conditioning regimen (if over 60 years old)
  * Melphalan 140 mg/m2 administered on Day -2 of transplant conditioning regimen.
  * Total Body Irradiation 2 Gray administered on Day -4, Day -3 of transplant conditioning regimen.
  * Tocilizumab 8 mg/kg administered on Day -1 of transplant conditioning regimen.
  Interventions: Drug: Tocilizumab; Drug: Fludarabine; Drug: Melphalan; Drug: Anti-thymocyte globulin (rabbit); Radiation: Total Body Irradiation
- ATG Group III (Experimental): Anti-thymocyte Globulin (ATG) 1.5 mg/kg administered on Day -5 of the transplant conditioning regimen.
  * Fludarabine 30mg/m2 administered on Day -7 through Day -3 of transplant conditioning regimen (if under 60 years old), or on Day -5 through Day -3 of transplant conditioning regimen (if over 60 years old)
  * Melphalan 140 mg/m2 administered on Day -2 of transplant conditioning regimen.
  * Total Body Irradiation 2 Gray administered on Day -4, Day -3 of transplant conditioning regimen.
  * Tocilizumab 8 mg/kg administered on Day -1 of transplant conditioning regimen.
  Interventions: Drug: Tocilizumab; Drug: Fludarabine; Drug: Melphalan; Drug: Anti-thymocyte globulin (rabbit); Radiation: Total Body Irradiation
- ATG Group IV (Experimental): * Fludarabine 30mg/m2 administered on Day -7 through Day -3 of transplant conditioning regimen (if under 60 years old), or on Day -5 through Day -3 of transplant conditioning regimen (if over 60 years old)
  * Melphalan 140 mg/m2 administered on Day -2 of transplant conditioning regimen.
  * Total Body Irradiation 2 Gray administered on Day -4, Day -3 of transplant conditioning regimen.
  * Tocilizumab 8 mg/kg administered on Day -1 of transplant conditioning regimen.
  Interventions: Drug: Tocilizumab; Drug: Fludarabine; Drug: Melphalan; Radiation: Total Body Irradiation

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab 8 mg/kg intravenously administered as a single dose on Day -1 of transplant conditioning regimen
  Other Names: Actemra
Drug: Fludarabine — Fludarabine 30 mg/m2 intravenously administered on Day -7, Day -6, Day -5, Day -4, Day -3 of transplant conditioning regimen if under the age of 60. If over the age of 60, Fludarabine 30 mg/m2 intravenously administered on Day -5, Day -4 and Day -3 of transplant conditioning regimen.
  Other Names: Fludara
Drug: Melphalan — Melphalan 140 mg/m2 intravenously administered on Day -2 of transplant conditioning regimen.
  Other Names: Alkeran
Drug: Anti-thymocyte globulin (rabbit) — Anti-thymocyte globulin (ATG) 1.5 mg/kg
  Other Names: Thymoglobulin
  Arms: ATG Group I; ATG Group II; ATG Group III
Radiation: Total Body Irradiation — Total Body Irradiation (TBI) 2 Gray, administered on Day -4 and Day -3 of transplant conditioning regimen

SUMMARY:
The purpose of this study is to evaluate the safety of reducing and ultimately eliminating anti-thymocyte globulin (ATG) from the haplo-cord transplant conditioning regimen and replacing it with tocilizumab, an IL-6 receptor monoclonal antibody, to improve immune reconstitution and reduce relapse while preserving low rates of graft failure and graft versus host disease (GVHD).

DETAILED DESCRIPTION:
This study is a prospective phase II non-inferiority study investigating tocilizumab as a potential alternative to anti-thymocyte globulin (ATG) in haplo-cord transplantation. It is a single-center study based at Weill Cornell Medicine/NewYork Presbyterian Hospital.

The hypothesis is that tocilizumab is a safe and effective alternative to ATG in haplo-cord transplantation, facilitating transient engraftment of the haplo-identical stem cell graft without prolonged neutropenia or second nadir prior to durable cord engraftment while also preventing graft versus host disease (GVHD).

This study plans to enroll patients with hematologic malignancies in need of alternate donor transplant. All subjects will be conditioned with fludarabine, melphalan and total body irradiation (TBI), followed by a single dose of tocilizumab 8 mg/kg on Day -1. Patients will be enrolled into 4 successive cohorts, initially administering the current standard 3 doses of ATG 1.5 mg/kg (total 4.5 mg/kg). In the absence of safety signals, we will drop one dose of ATG in successive cohorts until the drug ultimately has been eliminated.

The primary endpoint of the study is successful haplo-derived neutrophil engraftment. Treatment will only be of interest if there is evidence that this rate is greater than 60%. If there are 4 or fewer successes, that dose group will be deemed unacceptable and the next higher ATG dose for which there were 5 or more success will be expanded.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have a confirmed diagnosis of one of the following:

   1. Relapsed or refractory acute leukemia (myeloid or lymphoid)
   2. Acute leukemia in first remission at high-risk for recurrence
   3. Chronic myelogenous leukemia in chronic, accelerated phase or blast-crisis
   4. Myelodysplastic syndromes
   5. Chronic myeloproliferative disease
   6. Recurrent, refractory or high-risk malignant lymphoma
   7. Chronic lymphocytic leukemia, relapsed or with poor prognostic features
   8. Multiple myeloma
   9. Other hematological disorder in need of allogeneic transplant (e.g. blastoid dendritic cell neoplasm)
2. Age ≥ 18 years.
3. Likely to benefit from allogeneic transplant in the opinion of the transplant physician.
4. An HLA-identical related or unrelated donor cannot be identified within an appropriate time frame.
5. Karnofsky Performance Status (KPS) of ≥ 70%.
6. Acceptable organ function as defined below:

   1. Serum bilirubin: <2.0 mg/dL
   2. ALT (SGPT) <3x upper limit of normal (ULN)
   3. Creatinine Clearance: >50 mL/min/1.73m2 (eGFR as estimated by the modified MDRD equation)
   4. Left ventricular ejection fraction >40%
   5. Pulmonary diffusion capacity >40% predicted
7. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Life expectancy is severely limited by concomitant illness or uncontrolled infection.
2. Evidence of chronic active hepatitis or cirrhosis
3. Uncontrolled HIV disease.
4. Pregnancy or lactation.
5. History of complicated diverticulitis, including fistulae, abscess formation or gastrointestinal perforation
6. History of allergic reactions attributed to compounds of similar chemical or biological composition as tocilizumab, including known allergies to Chinese hamster ovary cell products or other recombinant human or humanized antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2027-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Gomez Arteaga, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ATG Group I: Anti-thymocyte Globulin (ATG) 1.5 mg/kg administered on Day -5, Day -3 and Day -1 of the transplant conditioning regimen.
  * Fludarabine 30mg/m2 administered on Day -7 through Day -3 of transplant conditioning regimen (if under 60 years old), or on Day -5 through Day -3 of transplant conditioning regimen (if over 60 years old)
  * Melphalan 140 mg/m2 administered on Day -2 of transplant conditioning regimen.
  * Total Body Irradiation 2 Gray administered on Day -4, Day -3 of transplant conditioning regimen.
  * Tocilizumab 8 mg/kg administered on Day -1 of transplant conditioning regimen.
  Tocilizumab: Tocilizumab 8 mg/kg intravenously administered as a single dose on Day -1 of transplant conditioning regimen
  Fludarabine: Fludarabine 30 mg/m2 intravenously administered on Day -7, Day -6, Day -5, Day -4, Day -3 of transplant conditioning regimen if under the age of 60. If over the age of 60, Fludarabine 30 mg/m2 intravenously administered on Day -5, Day -4 and Day -3 of transplant conditioning regimen.
  Melphalan: Melphalan 140 mg/m2 intravenously administered on Day -2 of transplant conditioning regimen.
  Anti-thymocyte globulin (rabbit): Anti-thymocyte globulin (ATG) 1.5 mg/kg
  Total Body Irradiation: Total Body Irradiation (TBI) 2 Gray, administered on Day -4 and Day -3 of transplant conditioning regimen
- ATG Group II: Anti-thymocyte Globulin (ATG) 1.5 mg/kg administered on Day -5, and Day -3 of the transplant conditioning regimen.
  * Fludarabine 30mg/m2 administered on Day -7 through Day -3 of transplant conditioning regimen (if under 60 years old), or on Day -5 through Day -3 of transplant conditioning regimen (if over 60 years old)
  * Melphalan 140 mg/m2 administered on Day -2 of transplant conditioning regimen.
  * Total Body Irradiation 2 Gray administered on Day -4, Day -3 of transplant conditioning regimen.
  * Tocilizumab 8 mg/kg administered on Day -1 of transplant conditioning regimen.
  Tocilizumab: Tocilizumab 8 mg/kg intravenously administered as a single dose on Day -1 of transplant conditioning regimen
  Fludarabine: Fludarabine 30 mg/m2 intravenously administered on Day -7, Day -6, Day -5, Day -4, Day -3 of transplant conditioning regimen if under the age of 60. If over the age of 60, Fludarabine 30 mg/m2 intravenously administered on Day -5, Day -4 and Day -3 of transplant conditioning regimen.
  Melphalan: Melphalan 140 mg/m2 intravenously administered on Day -2 of transplant conditioning regimen.
  Anti-thymocyte globulin (rabbit): Anti-thymocyte globulin (ATG) 1.5 mg/kg
  Total Body Irradiation: Total Body Irradiation (TBI) 2 Gray, administered on Day -4 and Day -3 of transplant conditioning regimen
- ATG Group III: Anti-thymocyte Globulin (ATG) 1.5 mg/kg administered on Day -5 of the transplant conditioning regimen.
  * Fludarabine 30mg/m2 administered on Day -7 through Day -3 of transplant conditioning regimen (if under 60 years old), or on Day -5 through Day -3 of transplant conditioning regimen (if over 60 years old)
  * Melphalan 140 mg/m2 administered on Day -2 of transplant conditioning regimen.
  * Total Body Irradiation 2 Gray administered on Day -4, Day -3 of transplant conditioning regimen.
  * Tocilizumab 8 mg/kg administered on Day -1 of transplant conditioning regimen.
  Tocilizumab: Tocilizumab 8 mg/kg intravenously administered as a single dose on Day -1 of transplant conditioning regimen
  Fludarabine: Fludarabine 30 mg/m2 intravenously administered on Day -7, Day -6, Day -5, Day -4, Day -3 of transplant conditioning regimen if under the age of 60. If over the age of 60, Fludarabine 30 mg/m2 intravenously administered on Day -5, Day -4 and Day -3 of transplant conditioning regimen.
  Melphalan: Melphalan 140 mg/m2 intravenously administered on Day -2 of transplant conditioning regimen.
  Anti-thymocyte globulin (rabbit): Anti-thymocyte globulin (ATG) 1.5 mg/kg
  Total Body Irradiation: Total Body Irradiation (TBI) 2 Gray, administered on Day -4 and Day -3 of transplant conditioning regimen
- ATG Group IV: * Fludarabine 30mg/m2 administered on Day -7 through Day -3 of transplant conditioning regimen (if under 60 years old), or on Day -5 through Day -3 of transplant conditioning regimen (if over 60 years old)
  * Melphalan 140 mg/m2 administered on Day -2 of transplant conditioning regimen.
  * Total Body Irradiation 2 Gray administered on Day -4, Day -3 of transplant conditioning regimen.
  * Tocilizumab 8 mg/kg administered on Day -1 of transplant conditioning regimen.
  Tocilizumab: Tocilizumab 8 mg/kg intravenously administered as a single dose on Day -1 of transplant conditioning regimen
  Fludarabine: Fludarabine 30 mg/m2 intravenously administered on Day -7, Day -6, Day -5, Day -4, Day -3 of transplant conditioning regimen if under the age of 60. If over the age of 60, Fludarabine 30 mg/m2 intravenously administered on Day -5, Day -4 and Day -3 of transplant conditioning regimen.
  Melphalan: Melphalan 140 mg/m2 intravenously administered on Day -2 of transplant conditioning regimen.
  Total Body Irradiation: Total Body Irradiation (TBI) 2 Gray, administered on Day -4 and Day -3 of transplant conditioning regimen
Period: Overall Study
Arm/Group | ATG Group I | ATG Group II | ATG Group III | ATG Group IV
Started | 10 | 10 | 1 | 0
Completed | 10 | 10 | 1 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No subjects were enrolled to ATG Group IV; study enrollment was stopped before accrual reached that cohort.
Groups:
- Total: Total of all reporting groups
Arm/Group | ATG Group I | ATG Group II | ATG Group III | ATG Group IV | Total
Number analyzed (Participants) | 10 | 10 | 1 | 0 | 21
Age, Customized [Count of Participants; unit: Participants]
  18-29 years | 1 | 2 | 0 | 0 | 3
  30-39 years | 1 | 2 | 0 | 0 | 3
  40-49 years | 1 | 2 | 0 | 0 | 3
  50-59 years | 0 | 1 | 0 | 0 | 1
  60-69 years | 7 | 3 | 1 | 0 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 1 | 0 | 11
  Male | 5 | 5 | 0 | 0 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 0 | 0 | 4
  Not Hispanic or Latino | 8 | 7 | 1 | 0 | 16
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 0 | 3
  White | 8 | 6 | 1 | 0 | 15
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 1 |  | 21
Primary Malignancy [Count of Participants; unit: Participants]
  Acute Myeloid Leukemia | 5 | 5 | 0 | 0 | 10
  Myelodysplastic Syndrome | 1 | 3 | 1 | 0 | 5
  Myeloproliferative Neoplasm | 1 | 1 | 0 | 0 | 2
  Non-Hodgkin Lymphoma | 2 | 1 | 0 | 0 | 3
  Other Acute Leukemia | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Successful Haplo-derived Neutrophil Engraftment
Description: This is defined as:
  1. Achieve an absolute neutrophil count (ANC) of 500 cells/microL for three consecutive days with the first on or prior to Day +21 post-transplant, AND
  2. Absence of a second nadir - a drop in the ANC to <300 cells/microL for five consecutive days - after initial neutrophil recovery.
Time Frame: 21 days post-transplant
Population: No subjects were enrolled to ATG Group IV; study enrollment was stopped before accrual reached that cohort.
Measure: Number; unit: percentage of participants
Arm/Group | ATG Group I | ATG Group II | ATG Group III | ATG Group IV
Number analyzed (Participants) | 10 | 10 | 1 | 0
percentage of participants | 80 | 50 | 0 |

2. Secondary Outcome: Progression-Free Survival
Description: Time elapsed between Day 0 and progression of the underlying malignancy for which the transplant was performed, assessed up to 5 years post-transplant.
Time Frame: 5 years post-transplant
Reporting Status: Not Posted

3. Secondary Outcome: Overall Survival
Description: Time elapsed between Day 0 and death from any cause, assessed up to 5 years post-transplant.
Time Frame: 5 years post-transplant
Reporting Status: Not Posted

4. Secondary Outcome: Transplant-Related Mortality
Description: Proportion of deaths which cannot be explained by persistence, relapse or progression of the underlying malignancy once the preparative regimen starts, assessed up to 5 years post-transplant.
Time Frame: 5 years post-transplant
Reporting Status: Not Posted

5. Secondary Outcome: Proportion of Platelet Engraftment Success
Description: Proportion of patients who successfully achieve platelet engraftment, defined as a platelet count of >20k/microL for three consecutive days without transfusion support for seven consecutive days.
Time Frame: 6 months post-transplant
Population: No subjects were enrolled to ATG Group IV, study enrollment was stopped before accrual reached that cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | ATG Group I | ATG Group II | ATG Group III | ATG Group IV
Number analyzed (Participants) | 10 | 10 | 1 | 0
Participants | 10 | 10 | 0 | 0

6. Secondary Outcome: Proportion of Failure of the Haplo-Graft
Description: Proportion of patients with a failed haplo-graft, defined as the absence of neutrophil engraftment by Day +21 or a drop in the absolute neutrophil count to <0.3 cells/microL for five consecutive days occurring after initial neutrophil engraftment within the first 3 weeks post-transplantation (second nadir)
Time Frame: 21 days post-transplant
Population: No subjects were enrolled to ATG Group IV; study enrollment was stopped before accrual reached that cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | ATG Group I | ATG Group II | ATG Group III | ATG Group IV
Number analyzed (Participants) | 10 | 10 | 1 | 0
Participants | 2 | 5 | 1 |

7. Secondary Outcome: Proportion of Acute Graft-versus-Host Disease
Description: Proportion of patients who develop acute graft-versus-host disease
Time Frame: 1 year post-transplant
Population: No subjects were enrolled to ATG Group IV, study enrollment was stopped before accrual reached that cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | ATG Group I | ATG Group II | ATG Group III | ATG Group IV
Number analyzed (Participants) | 10 | 10 | 1 | 0
Participants | 2 | 1 | 1 | 0

8. Secondary Outcome: Percentage of Chronic Graft-versus-Host Disease
Description: Percentage of patients who develop chronic graft-versus-host disease
Time Frame: 5 years post-transplant
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All-cause mortality is being assessed up to 5 years. SAEs and other non-serious AEs were assessed up to 1 year.
Description: No subjects were enrolled to ATG Group IV; study enrollment was stopped before accrual reached that cohort.
Arm/Group | ATG Group I | ATG Group II | ATG Group III | ATG Group IV
All-Cause Mortality (participants affected / at risk) | 5/10 | 1/10 | 1/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 8/10 | 9/10 | 1/1 | 0/0
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 1/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATG Group I (N=10) | ATG Group II (N=10) | ATG Group III (N=1) | ATG Group IV (N=0)
Acute Graft-versus-Host Disease (Investigations) | 1 (1) | 0 (0) | 1 (1) | NA
Bacteremia (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | NA
Hemophagocytic lymphohistiocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | NA
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | NA
Colitis - Cytomegalovirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | NA
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | NA
Delayed Engraftment (Investigations) | 0 (0) | 0 (0) | 1 (1) | NA
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | NA
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | NA
Failure to Thrive (General disorders) | 1 (1) | 1 (1) | 0 (0) | NA
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | NA
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | NA
Hypovolemic shock (General disorders) | 0 (0) | 0 (0) | 1 (1) | NA
Hemolytic Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | NA
Herpes simplex Reactivation (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | NA
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | NA
Lung Infection - COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | NA
Lung Infection -Chlamydia trachomatis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | NA
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | NA
Pancreatic Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | NA
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | NA
Sepsis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | NA
Septic Shock (Investigations) | 2 (3) | 1 (1) | 1 (1) | NA
Sinusoidal Obstruction Syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | NA
Throat Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | NA
Upper Respiratory Infection - Coronavirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | NA
Upper Respiratory Infection - Human Metapneumovirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | NA
Upper Respiratory Infection - Parainfluenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | NA
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | NA
Viremia - Cytomegalovirus (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATG Group I (N=10) | ATG Group II (N=10) | ATG Group III (N=1) | ATG Group IV (N=0)
Acute Graft-versus-Host Disease (Investigations) | 3 (3) | 2 (2) | 0 (0) | 0
Viremia - Adenovirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0
Adenovirus Colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0
Alanine aminotransferase increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0
Anemia (Blood and lymphatic system disorders) | 9 (9) | 10 (10) | 1 (1) | 0
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 0 (0) | NA
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1) | 0 (0) | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 1 (1) | 0
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 1 (1) | 0
Hypokalemia (Metabolism and nutrition disorders) | 4 (4) | 4 (4) | 1 (1) | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1) | 0
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0
Platelet count decreased (Investigations) | 6 (6) | 4 (4) | 1 (1) | 0
White blood cell decreased (Investigations) | 1 (1) | 3 (3) | 1 (1) | 0
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (3) | 0 (0) | 0
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 0
Upper Respiratory Infection - Parainfluenza (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0
Upper Respiratory Infection - Rhinovirus (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0
Upper Respiratory Infection - Coronavirus (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0
Upper Respiratory Infection - COVID-19 (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0
Viremia - Cytomegalovirus (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0
Upper Respiratory Infection - Respiratory Syncytial Virus (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0
Hemolytic Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0
Bacteremia (Infections and infestations) | 2 (2) | 3 (3) | 1 (1) | 0
Infectious Colitis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0
Candida pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0
BK Virus Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT04395222/Prot_SAP_000.pdf